CLINICAL TRIAL: NCT05811650
Title: Effect of School-based Oral Health Promotion and Counselling Interventions Among School Children in Nepal: A Cluster Randomized Controlled Trial
Brief Title: School Oral Health Intervention in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyberjaya University College of Medical Sciences (Other)
Responsible Party: Principal Investigator, Kamal Prasad Chapain, PhD scholar, Cyberjaya University College of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNP-1-PHD-1901001
Record Dates: First submitted 2023-03-11; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: The intervention will target school teachers and school children for counseling and oral health promotion education
Who Masked: Participant
Masking Description: School Children in the control group will be in control and will not receive any intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Health Intervention group (Experimental): Those receiving intervention of oral health and counselling.
  Interventions: Behavioral: Oral Health Counseling and promotion
- Control group (Placebo Comparator): Those who are not receiving counseling and promotion interventions
  Interventions: Behavioral: Oral Health Counseling and promotion

INTERVENTIONS:
Behavioral: Oral Health Counseling and promotion — The intervention was cluster randomized control trial in design. We select six schools for the intervention group and six schools for the control group. Follow-up of the intervention was done after six months of baseline. Impact of the intervention was assessed among the same participants who enrolled in the baseline. The interventions were done in every three months.

SUMMARY:
Oral health problems in school children are highly prevalent in Nepal. The investigators designed oral health counseling and promotion intervention in Kaski district of Nepal for six months. The study was conducted intervention covering dental check up, counseling, supporting with brush materials, toothpaste, and essentials. The investigators also trained school teachers to provide oral health education in school children and completed the endline data collection to assess the effect of intervention.

DETAILED DESCRIPTION:
Globally oral health diseases are common health problems in children. About 60-90% of school children are suffering from dental caries worldwide . Dental caries is the most prevalent condition included in the 2016 Global Burden of Disease Study, ranking the first for the decay of permanent teeth (2.3 billon people) and 12th for deciduous teeth (560 million children). The dental caries process begins with a small patch of demineralized (softened) enamel at the tooth surface and the destruction then spreads into the softer, sensitive part of the tooth beneath enamel (dentin).

Common oral diseases among children are dental caries and periodontal diseases . Pain from teeth or mouth can compromise their concentration and their participation in school, thereby hampering not only their play and development but also denying them the full benefit of schooling. In addition, such oral health problems negatively affect a child in restricting their activities, reducing the ability to learn, and increasing the frequency of absenteeism from schools . The most common cause of the dental problem is due to lack of dental health education, negligence of treatment in an early stage. Children do not have the knowledge to choose proper toothpaste and brush which plays an important role to maintain their oral hygiene and prevention dental caries. To improve oral health conditions proper awareness level plays an important role. Also, the proper method of tooth brushing plays an important role to maintain oral health status.

A national Pathfinder Survey. However, there is no evidence in higher grade children in schools. The problem is grave in school children and little or no interventions targeting children have been practiced in Nepal.

Therefore, designing an effective intervention that addresses knowledge and behavior on oral health targeting school children is necessary because they are the most at-risk population of oral health problems in Nepal and elsewhere. The overall aim of this study is to assess the effect of oral health promotion and counseling interventions on knowledge and oral hygiene practices in school children in Pokhara, Nepal.

A cluster randomized control trial study will be conducted in selected community schools of Kaski District of Nepal. We will select six schools for the intervention group and six schools for the control group. The study sample will be the school students in the selected schools of 7 and 8 Grades. The sampling frame will be determined after preparing the list of students totaling of 580 students (Intervention:290; Control:290). The investigator will measure students' demographic characteristics, knowledge, and practices in oral health. The study will be conducted one year of an intervention comprising oral health screening and counseling every three months in the intervention group and will examine the effect of school-based intervention after one year of intervention. This study is expected to provide evidence to develop strategies for oral health promotion in community schools in Nepal.

ELIGIBILITY:
Inclusion Criteria

* The school children, who have studied in the schools at least one year before the start of the study.
* Grade 7

Exclusion Criteria:

- The school children, who were absent for more than one week before the start of the study

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 669 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
DMFT index | 6 months
  The is the index developed by WHO. DMFT is the sum of the number of Decayed, Missing due to caries, and Filled Teeth in the permanent teeth. The highest score is 32 and lowest is zero
Oral Health Knowledge | 6 months
  The total oral health knowledge score was ranging from 0-9 being nine as the highest score. The response of the knowledge test was measures as: Yes = 1, No and Don't Know = 0.
Practice on oral health | 6 month
  Prevalence of children who had better practices of health. Proportion of those who have regular tooth brushing, mouth gargle, tongue cleaning, and dental flush
Health Seeking Behavior | 6 monhts
  Proportion of people who have improved health seeking behavior in intervention compared to control

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kamal Pr Chapain, BDS, MPH, Principal Investigator — Paschimanchal Dental Home
Locations (1):
- Paschimanchal Dental Home, Pokhara, Gandaki, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with genuine request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after the completion of the study
Access Criteria: Request with email to PI